CLINICAL TRIAL: NCT04802525
Title: A Low-fat Diet Combined With Moderate-intensity Aerobic Exercise is More Effective Than a Low-fat Diet or Aerobic Exercise Alone on Dyslipidemia and Depression Status in Obese Patients
Brief Title: A Low-fat Diet Combined With Moderate-intensity Aerobic Exercise Versus Low-fat Diet, Aerobic Exercise Alone on Dyslipidemia and Depression Status in Obese Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Marwa Eid, assistant professor of physical therapy for surgery, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: obesity 2
Record Dates: First submitted 2021-03-15; First posted 2021-03-17 (Actual); Last update posted 2021-03-17 (Actual); Status verified 2021-03

CONDITIONS: Dyslipidemias
MeSH Terms: conditions — Dyslipidemias

STUDY DESIGN:
Who Masked: Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Moderate-intensity aerobic exercise training without dietary control group (Experimental)
  Interventions: Other: Moderate-intensity aerobic exercise training
- Low-fat diet program without exercise intervention group (Experimental)
  Interventions: Other: Moderate-intensity aerobic exercise training
- Moderate-intensity aerobic exercise training plus a low-fat diet program group (Experimental)
  Interventions: Other: Moderate-intensity aerobic exercise training

INTERVENTIONS:
Other: Moderate-intensity aerobic exercise training — The first group has received Moderate-intensity aerobic exercise training without dietary control, the second group has received a low-fat diet program without exercise intervention, and the third group has received Moderate-intensity aerobic exercise training plus a low-fat diet program for 10 consecutive weeks

SUMMARY:
It was defined that exercise and dietary interventions are used to control dyslipidemia and depression in obese individuals, whilst rare investigations have examined the concurrent effects of a low-fat diet and moderate-intensity aerobic exercise training (MIAET) on dyslipidemia and depression in obese patients. Hence, we assessed the potential influences of a low-fat diet combined with MIAET on blood lipids and depression in those individuals.

ELIGIBILITY:
Inclusion Criteria:

* age of 30-50 years
* clinical diagnosis with obesity (BMI˃30)
* mild to moderate depression
* impaired blood lipids
* no use of medications last 6-12 months
* no smoking

Exclusion Criteria:

* neuromuscular, endocrinal, musculoskeletal, cardiovascular disorders
* severe depression
* patients using medications of dyslipidemia, depression, or obesity last 6-12 months.

Ages: 30 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 42 (Actual)
Dates: Start 2019-10-10 (Actual); Primary Completion 2020-01-02 (Actual); Study Completion 2020-01-15 (Actual)

PRIMARY OUTCOMES:
Body Mass Index | 10 weeks
  The height and weight were assessed using an electronic digital scale and consequently BMI was calculated

CONTACTS AND LOCATIONS:
Locations (1):
- Marwa Eid, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No